CLINICAL TRIAL: NCT01484665
Title: Evaluating the Effect of a Decision Aid on Shared Decision Making for Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2011NTLS071
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer
Keywords: PSA screening; Decision aids
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants (Males, age 50-75 yrs) (Experimental): Eligible men will be identified from the administrative database and electronic medical record at the University of Minnesota (EMR) at least 24 hours prior to the clinic visit. They will be asked to complete the PROCASE Decision-Aid.
  Interventions: Other: PROCASE Decision-Aid

INTERVENTIONS:
Other: PROCASE Decision-Aid — VA health services researchers have developed a patient education pamphlet for prostate cancer screening. The pamphlet, titled "The PSA test for prostate cancer: Is it Right for ME was created by members of the PROstate CAncer Screening Education (PROCASE) study team. A modified version of the PROCASE decision aid will be utilized in this study.

SUMMARY:
Decision-aids are tools to educate patients on a given topic so that they may better participate in shared-decision making in their health care. Given the complexities associated with PSA testing, many professional organizations have advocated for shared-decision making for PSA testing. However, no consensus exists as to how best educate and involve patients in the shared-decision making process. The goal of this study is to evaluate a pilot program utilizing a simple PSA screening decision-aid presented in two different fashions in a primary care clinic with a large fraction of African-American patients. The investigators will evaluate the effectiveness of this program to educate patients on the risks and benefits of prostate specific antigen (PSA) testing, on their subsequent level of comfort with their decision about whether to receive PSA testing, and on the comfort level of physicians on their patient's decisions regarding PSA testing, and importantly, how well these strategies can be implemented into the daily work-flow of a clinic. If successful, this program may serve as a model for the broader implementation of such strategies across Minnesota and the country.

DETAILED DESCRIPTION:
This pilot project will evaluate two approaches to implementing the use of a simple printed PSA screening decision-aid (DA) administered in an urban primary care clinic populated with a significant number of African-Americans. All subjects will complete a survey assessing their knowledge and attitudes about PSA screening and shared decision making (SDM), and physicians will also be briefly queried about their perceptions of the SDM process.

After the first three month implementation period we will conduct focus groups with clinic staff to guide changes and refinements to the use of DA in the clinical setting. Another three month implementation period will follow using the same methods to assess outcomes. Finally we will conduct another round of focus groups to assess the overall impact of the interventions.

ELIGIBILITY:
Inclusion criteria:

* Males ages 50-75
* Able to read and speak English
* Provide written informed consent

Exclusion criteria:

* Diagnosis of prostate cancer
* PSA testing within last 12 months
* Previous prostate biopsy
* Voiding problems as reason for clinic visit
* Visit scheduled same day or 'walk-In' patient

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Provider Satisfaction with Implementation of the Shared Decision Making Process | At 3-5 Months
  Will be determined through a combination of surveys and responses to questions derived during focus groups.
Provider Satisfaction with Implementation of the Shared Decision Making Process | At 8-10 Months
  Will be determined through a combination of surveys and responses to questions derived during focus groups.

SECONDARY OUTCOMES:
Patient Satisfaction with Shared Decision Making and Reach of the Intervention | At 8-10 Months
  Will be determined through a questionnaire administered to patients.
Patient Satisfaction with Shared Decision Making and Reach of the Intervention | At 3-5 Months
  Will be determined through a questionnaire administered to patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Warlick, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Broadway Family Medicine Clinic, Minneapolis, Minnesota, United States